CLINICAL TRIAL: NCT02804113
Title: VMI-CFA Study: Physician-initiated Trial Investigating the Efficacy of the Vascular Mimetic Implant Supera Peripheral Stent System for the Treatment of the Common Femoral Artery
Brief Title: Clinical Trial Investigating the Efficacy of the Supera Peripheral Stent System for the Treatment of the Common Femoral Artery
Acronym: VMI-CFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ID3 Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iD3 Medical - 160226
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

ARMS (1):
- Supera Peripheral Stent System (Experimental)
  Interventions: Device: Supera Peripheral Stent System

INTERVENTIONS:
Device: Supera Peripheral Stent System

SUMMARY:
The VMI-CFA study investigates the efficacy of the Supera Stent in the treatment of common femoral artery stenosis or occlusion. 100 patients will be included with a RF of 2 to 4. The lesion is located within the native CFA and treated with predillation prior to stenting with the Supera Peripheral Stent System. Patients will be invited for a follow-up visit at 1, 6, 12 and 24 month post procedure. The primary endpoint of the study is the primary patency at 12 months and periprocedural events up to 30 days post procedure. Secondary endpoints include technical success, primary patency rate at 1, 6 and 24 month, freedom from TLR at 1-, 6-, 12 and 24 month follow-up and clinical success at 1-, 6-, 12- and 24-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting a score from 2 to 4 following Rutherford classification
* Patient is willing to comply with specified follow-up evaluations at the specified times
* Patient is >18 years old
* Patient understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
* Patient has a projected life expectancy of at least 12 months
* Prior to enrolment, the guidewire has crossed target lesion
* De novo lesions located in the common femoral artery, suitable for endovascular therapy
* The target lesions are located within the native CFA: localized between the origin of the circumflex iliac artery and the proximal (1cm) superficial femoral artery.
* There is angiographic evidence of a patent deep femoral artery
* The target lesion has angiographic evidence of stenosis > 50% or occlusion
* There is angiographic evidence of at least one-vessel-runoff to the foot, irrespective of whether or not outflow was re-established by means of previous endovascular intervention

Exclusion Criteria:

* Presence of another stent in the target vessel that was placed during a previous procedure
* Previous open surgery in the same limb
* Patients contraindicated for antiplatelet therapy, anticoagulants or thrombolytics.
* Patients who exhibit persistent acute intraluminal thrombus at the target lesion site.
* Perforation at the angioplasty site evidenced by extravasation of contrast medium
* Patients with known hypersensitivity to nickel-titanium and heparin, including those patients who have had a previous incidence of heparin-induced thrombocytopenia (HIT) type II
* Patients with uncorrected bleeding disorders
* Female patient with child bearing potential not taking adequate contraceptives or currently breastfeeding
* Ipsilateral inflow (aorto-iliac) artery treatment before target lesion treatment with a residual stenosis>30%
* Use of thrombectomy, atherectomy or laser devices during procedure
* Any planned surgical intervention/procedure 30 days after the study procedure
* Any patient considered to be hemodynamically unstable at onset of procedure
* Patient is currently participating in another investigational drug or device study that has not reached the primary endpoint.
* Severe medical comorbidities (untreated CAD/CHF, severe COPD, metastatic malignancy, dementia, etc.) or other medical condition that would preclude compliance with the study protocol or 1-year life expectancy
* Major distal amputation (above the transmetatarsal) in the study limb or non-study limb
* Septicemia or bacteremia
* Known allergy to contrast media that cannot be adequately pre-medicated prior to the study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Primary patency at 12 months | 12 months
  freedom from > 50% restenosis as indicated by an independently verified duplex ultrasound peak systolic velocity ratio (PSVR) <2.5 in the target vessel with no reintervention (TLR) within 12 months.
Periprocedural adverse events | 30 days post procedure
  periprocedural adverse events up to 30 days post procedure, as defined per ISO 14155:2011

SECONDARY OUTCOMES:
Technical success | during indexprocedure
  ability to cross and stent the lesion to achieve residual angiographic stenosis no greater than 30% and residual stenosis less than 50% by duplex imaging.
Primary patency rate at 1, 6 and 24 month | 1, 6 and 24 month post procedure
  freedom from >50% restenosis as indicated by an independently verified duplex ultrasound peak systolic velocity ratio (PSVR) <2.5 in the target vessel with no intervention within 1 and 6 months.
Freedom from TLR until 24 month post procedure | until 24 month post procedure
  freedom from a repeat intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5mm proximal and distal to the treated lesion edge at the respective time points
Clinical success | 1, 6, 12 and 24 month follow-up
  an improvement of Rutherford classification at 1-, 6-, 12- and 24-month follow-up of one class or more as compared to the pre-procedure Rutherford classification.

CONTACTS AND LOCATIONS:
Overall Officials: Koen Deloose, MD, Study Director — ID3 Medical
Locations (7):
- Belgium (4):
  - ZNA Stuivenberg, Antwerp, Antwerp
  - OLV Ziekenhuis Aalst, Aalst, Oost-Vlaanderen
  - AZ Sint-Blasius, Dendermonde, Oost-Vlaanderen
  - Imelda Hospital, Bonheiden
- France (3):
  - Clinique Rhone Durance, Avignon
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Nantes, Nantes